CLINICAL TRIAL: NCT06334016
Title: Acute Effects of Sequential Nicotine Vaping on the Pharmacokinetic and Pharmacodynamic Properties of Vaped THC: A Double-Blind, Placebo-Controlled, Randomized Within-Subject Crossover Study
Brief Title: Evaluating the Delivery and Effects of THC Vaping Liquids in the Bloodstream
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: I-3597023; NCI-2024-01556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3597023 (Other: Roswell Park Cancer Institute); R01DA057228 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Specimen Handling; nabiximols; Nicotine

STUDY DESIGN:
Intervention Model Description: Within-subject crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and clinical personnel will be blinded to the nicotine product sequence (active vs. placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (placebo, THC, nicotine) (Experimental): Participants complete 3 vaping sessions separated by 7-14 days on study:
  * VISIT 1: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.
  * VISIT 2: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.
  * VISIT 3: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.
  All participants also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cannabis sativa Extract; Drug: Nicotine; Drug: Placebo Administration; Other: Questionnaire Administration
- Arm B (placebo, THC, nicotine) (Experimental): Participants complete 3 vaping sessions separated by 7-14 days on study:
  * VISIT 1: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.
  * VISIT 2: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.
  * VISIT 3: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.
  All participants also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cannabis sativa Extract; Drug: Nicotine; Drug: Placebo Administration; Other: Questionnaire Administration
- Arm C (placebo, THC, nicotine) (Experimental): Participants complete 3 vaping sessions separated by 7-14 days on study:
  * VISIT 1: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.
  * VISIT 2: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.
  * VISIT 3: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.
  All participants also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cannabis sativa Extract; Drug: Nicotine; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cannabis sativa Extract — Vape THC
  Other Names: Cannabis sativa; Cannabis sativa Flowering Top; Cannabis sativa Subsp. Flowering Top Extract; Cannabis sativa Top
Drug: Nicotine — Vape active nicotine
  Other Names: (-)-Nicotine; NIC
Drug: Placebo Administration — Vape placebo nicotine
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial assesses differences in the delivery of THC to the bloodstream depending on whether nicotine vapes are used before or after THC. While there has been much recent publicity about vaping products and concern about their safety considering their increasing use for THC administration, the THC delivery profile associated with THC liquid vaping products in human subjects is currently unknown. Importantly, how the delivery to the bloodstream of THC vaping liquids compare to delivery from smoked cannabis, which is the most used method of cannabis delivery, will serve as an important benchmark for evaluating the delivery and effects of THC vaping products, and their relative safety.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess pharmacokinetic (PK)/pharmacodynamic (PD) profiles of THC vaping liquids administered with co-use of vaped nicotine.

II. Outcomes of interest will be assessed overall, and according to biological sex.

SECONDARY OBJECTIVES:

I. Safety. II. Assessment of differences in puffing behaviors. III. Short-term subjective drug effects, and cognitive performance following THC use without nicotine versus (vs.) THC use with pre-nicotine use vs. THC use with post-nicotine use in current consumers of both vaped cannabis and vaped nicotine products.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM A: Participants complete 3 vaping sessions separated by 7-14 days on study:

* VISIT 1: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.
* VISIT 2: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.
* VISIT 3: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.

ARM B: Participants complete 3 vaping sessions separated by 7-14 days on study:

* VISIT 1: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.
* VISIT 2: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.
* VISIT 3: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.

ARM C: Participants complete 3 vaping sessions separated by 7-14 days on study:

* VISIT 1: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then nicotine for 10 minutes.
* VISIT 2: Participants vape placebo nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine again for 10 minutes.
* VISIT 3: Participants vape nicotine for 10 minutes, followed by THC for 10 minutes, and then placebo nicotine for 10 minutes.

All participants also undergo blood sample collection throughout the trial.

After completion of study intervention, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years of age; (self-reported on screening, verified at study visit).
* Report use of commercial THC vaping cartridges for at least 3 months prior to enrollment; (self-reported).
* Experience with THC potency at or above the study product AND experience with chasing THC with nicotine (at least monthly); (self-reported).
* Report use of THC vaping liquids at least weekly (4x/month); (self-reported).
* Daily use of nicotine vaping products containing 5% nicotine for at least 3 months prior to enrollment; (self-reported).
* Report of not currently trying to become pregnant (females). Women of childbearing potential must be willing to provide a urine sample and test negative prior to receiving any study-related products/procedures.
* Willing to complete a THC saliva test to check for recent use (NarcoCheck Ref#: NCE-STHC-1), semi-quantitative urinary THCA rapid test (NarcoCheck® THC Pre Dosage), and an illicit drug urine test (NarcoCheck® Évolutive®) during baseline testing, prior to receiving any study-related products.
* Negative THC saliva test (NarcoCheck Ref#: NCE-S-THC-1), detection level 1-3 on urinary THCA rapid test (NarcoCheck® THC PreDosage), and illicit drug screen negative for all drugs except THC (NarcoCheck® Évolutive®).
* Willing to abstain from nicotine use for 8 hours prior to each study session and abstain from cannabis use 7 days prior to each session.
* Participant must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Detection level 4-5 (> 300 ng/mL) on urinary THCA rapid test (NarcoCheck® THC PreDosage Ref#: DOA-M03-9B) and a positive result on THC saliva test (NarcoCheck Ref#: NCE-S-THC-1).
* Illegal or non-prescription drug use within the past 90 days. As detected by NarcoCheck® Évolutive® (detection in human urine of the 12 most currently abused drugs) at the first session and prior to receiving any study product. THC use detected by NarcoCheck® Évolutive® is permitted
* Illegal or non-prescription drug use/alcohol substance use disorder (SUD) within the past year; (self-reported).
* Report 2 or more drinking occasions/week with 4 or more drinks/occasion; (self-reported).
* Report of daily cigarette use; (self-reported).
* Current or prior diagnosis of schizophrenia, bipolar disorder, or other severe psychotic mental illness; (self-reported).
* Current or prior diagnosis of myocardial infarction, arrhythmia, or congestive heart failure (self-reported).
* Current or prior cancer diagnosis.
* Pregnant, currently trying to become pregnant, or breastfeeding (females); (self-reported; pregnancy validated on study visit by urine test).
* Regular use of medications that contain nicotine, induce CYP2A6, stimulants, or sympatholytics (e.g., beta-blockers); (self-reported).
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate for participation.
* The following special populations will be excluded:

  * Cognitively impaired adults/adults with impaired decision-making capacity
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners
* No children or person under the age of 21 will be involved in the study. While those under 21 may use cannabis smoked or vaping products, the legal age of purchasing and using those products in New York State is 21. The current legal age to purchase and use tobacco products in New York State (NYS) is 21. Thus, our provision of study product to adults aged 21 and older is in line with current NYS law.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of THC in plasma (Cmax) | Up to 21 days
  Pharmacokinetics (PK) profiles of THC in plasma will be determined using a visual plot of plasma THC concentrations by time. Parameters will be derived using non-compartmental analysis in Phoenix WinNonlin and adjusted for baseline THC levels. Will be summarized by nicotine status using the appropriate descriptive statistics and graphical summaries.
Area under the plasma concentration-time curve from 0-360 minutes (AUC0-360) | Up to 21 days
  Blood samples will be collected for plasma levels of THC. Parameters will be derived using linear mixed models
Time to maximum concentration of THC in plasma (Tmax) | Up to 21 days
  Blood samples will be collected for plasma levels of THC. Parameters will be derived using linear mixed models.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after completion of study intervention
  AEs will be summarized by nicotine condition and grade using frequencies and relative frequencies. Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.
Puffing behaviors | Up to 21 days
  puff duration
Puffing behaviors | Up to 21 days
  puff number
Short-term drug effects | Up to 21 days
  The short-term drug effects (Drug Effects Questionnaire [DEQ), The DEQ rates sixteen component items using a visual analog scale (0-100) to examine drug effects pre- and post-use
Marijuana Withdrawal Checklist [MWC) | Up to 21 days
  The Marijuana Withdrawal Questionnaire Total Score includes items assessing anxiety, depression, irritability, appetite, aggression/anger, sleep disturbance, somatic disturbances, and craving to use marijuana. The potential range of this total score is from "0" = no withdrawal symptoms to "47" = maximally high levels of withdrawal
Digit Symbol Substitution Task (DSST) | Up to 21 days
  An assessment of cognitive dysfunction that test ability to complete daily tasks
Paced Auditory Serial Addition Task (PASET) | Up to 21 days
  Measures of working memory and concentration .
Tobacco Craving Questionnaire (Short Form) | Up to 21 days
  Self reported 47-item questionnaire that assesses tobacco craving. Items are rated on a Likert-type scale from 1 (strongly disagree) to 7 (strongly agree). Factor scores for each participant are obtained by summing the three items in each factor scale, yielding a score ranging from 3 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Smith, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States